CLINICAL TRIAL: NCT02583555
Title: Randomised Case Management Study to Reduce Health Care Utilization for Frequent Hospital Care Users
Brief Title: Case Management Study to Reduce Health Care Utilization for Frequent Hospital Care Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Sjælland (Other)
Collaborators: Health Navigator (Other)
Responsible Party: Principal Investigator, Knud Rasmussen, MD, DMSci, Research Consultant, MD, DMSci, Region Sjælland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJ-499
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Quality of Life
Keywords: Quality of Life; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active patient support (Active Comparator): Interview followed by frequent telephone support Questionnaire every 3 months
  Interventions: Behavioral: Interview followed by frequent telephone support
- Controls (No Intervention): Questionnaire every 3 months

INTERVENTIONS:
Behavioral: Interview followed by frequent telephone support — Interview followed by telephone support
  Arms: Active patient support

SUMMARY:
The purpose of this study is to identify persons with high risk of frequent hospital admissions and by counselling by one in depth interview followed by frequent telephone contacts improve their quality of life and reduce their healthcare utilization.

DETAILED DESCRIPTION:
Participants are identified by administrative data and a model predicting high risk of future healthcare utilization. Participants are invited to the study by mail. After informed consent participants are randomized to either active treatment or control 3:1. Active patients have an in depth interview with a specially trained nurse. Further counselling by telephone weekly for 6-9 months.

Quality of Life is measured by SF-36 every 3 months for one year both in active participants and in controls.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years
* Recent history of contact with hospital
* Anticipated sustained high visit frequency

Exclusion Criteria:

* Dementia (ICD10: F00-F03 or F051)
* Psychoses (ICD10: F20-F29)
* Drug abuse (ICD10: F10-F19)
* Metastases (ICD10: C77-C80)
* Hearing impairment or language difficulties
* Life expectancy < 1 year No telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life reported by the participants with use of Short Form 36 | Questionaire Short Form-36 Every 3 months for one year
Health Care Utilization - Admissions to and days in hospital | One year
  The use of different health care systems will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Knud Rasmussen, MD DMSci, Principal Investigator — Research Consultant
Locations (1):
- Regional Research, Roskilde, Denmark